CLINICAL TRIAL: NCT02812017
Title: Thirty Million Words: Well Baby Initiative
Brief Title: Thirty Million Words- Well Baby Initiative
Acronym: TMW-WB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 15-0914
Record Dates: First submitted 2016-06-22; First posted 2016-06-23 (Estimated); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Behavior; Communication; Language
Keywords: educational intervention; language development; postpartum; parental attachment; achievement gap; language gap; school readiness
MeSH Terms: conditions — Behavior; Communication; Language

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 - Intervention (Experimental): The treatment group will complete a demographics questionnaire and the baseline measures before the intervention. Participants will then view the Thirty Million Words-Well Baby intervention, which consists of educational, multimedia modules at the one-, two-, four-, and six-month well baby pediatric visits. The participant will complete survey measures after the one-, two-, four- and six-month visits, as well as over email at seven-months old and in clinic again at the nine-, twelve-, eighteen-, and twenty-four month visits.
  Interventions: Behavioral: Thirty Million Words- Well Baby
- 2 - Neutral (Placebo Comparator): The Neutral Video group will complete a demographics questionnaire and the baseline measures before the intervention. Participants will then view the neutral videos about car safety at the one-, two-, four-, and six-month well baby pediatric visits. The participant will complete survey measures after the one-, two-, four- and six-month visits, as well as over email at seven-months old and in clinic again at the nine-, twelve-, eighteen-, and twenty-four month visits.
  Interventions: Other: Safety Starts at Home
- 3 - Usual care (No Intervention): The treatment group will complete a demographics questionnaire and the baseline measures before the intervention. Participants will receive care as usual at the one-, two-, four-, and six-month well baby pediatric visits. The participant will complete survey measures after the one-, two-, four- and six-month visits, as well as over email at seven-months old and in clinic again at the nine-, twelve-, eighteen-, and twenty-four month visits.

INTERVENTIONS:
Behavioral: Thirty Million Words- Well Baby — Through evidence-based strategies, the TMW-WB curriculum teaches parents how to harness the power of their words to build their child's brain and impact their child's learning trajectory.
  Arms: 1 - Intervention
Other: Safety Starts at Home — A portion of the Safety Stars at Home set is shown. Demonstrating proven childproofing techniques and accident-prevention strategies, which unifies safety guidelines and shows caregivers how to take proactive measures at home. Many no- or low-cost safety alternatives are offered.
  Arms: 2 - Neutral

SUMMARY:
The purpose of the proposed study is to determine the efficacy of a multi-media educational curriculum in strengthening the early learning environments of vulnerable children, and positively impacting their language and cognitive development. Through evidence-based strategies, the TMW-WB curriculum teaches parents how to harness the power of their words to build their child's brain and impact their child's learning trajectory.

DETAILED DESCRIPTION:
Participants will be recruited at Lawndale Christian Health Clinic (LCHC), Advocate Medical Group (AMG), or PCC Community Wellness Centers (PCC) at their first well-baby visit. If the parent and child are eligible for the study, the parents will be asked to give informed consent for the study.

Before the one-month visit, participants will be randomized into the three experiential groups. We will use the website Research Randomizer to generate a randomization table. We will use the service to generate a dummy set of 500 unique unsorted numbers where each unique number is paired with a participant number (1-250, sorted). In an Excel spreadsheet, the first half of the dummy number set) will be assigned evenly to the Treatment condition (arm 1) and the other half will be assigned evenly to the Control conditions (arms 2 or 3). Then, the data in the columns "participant", "condition" and "dummy" will be sorted using the Excel "Sort by" function on the column "dummy". The participant numbers are now unsorted and randomly assigned to either one of the two experimental conditions: Treatment or Control. The treatment group will be randomized again in the same way as explained above to either TMW-Well Baby arm, orthe two control groups Usual Care arm Neutral Video arm. This will allow us to ensure equal sample sizes for all treatment and control conditions. A separate randomization table will be crated in the same way for the Spanish-speaking group.

At the one-month Well Baby visit, participants in the Usual Care arm of the study will receive care as usual. Participants in the Neutral Video arm will watch the first of four short videos (approximately 5-10 minutes) about infant safety. Patients in the TMW-Well Baby arm will watch the Module 1 video intervention. This module present information on child language and cognitive development. Videos will be shown in the waiting room, or during the period after the nurse completes the child's vitals and before the pediatrician sees the patient. Should a video still be running when the pediatrician enters the room, it will be stopped and completed after the pediatrician has left. After the visit, patients in all arms will be asked to complete the Post-Visit survey about their visit, indicating the areas and level of anticipatory guidance they received during their visit, their overall satisfaction levels, and their unmet needs for guidance and requests for more information. At this visit, the health clinic may collect information using a standardized depression scale. This provides information on the covariates parental language ability and depression level. Results from the depression scale will be shared by the patient's pediatrician, both because pediatricians need to administer a depression scale anyway and in an effort to reduce burdens associated with housing the study in the clinic. If the clinic does not administer a depression scale, the Edinburgh Postnatal Depression Scale (EPDS)will be administered by the research staff.

At their two-month Well Baby visit, patients in the TMW-Well Baby arms will watch the Module 2 video intervention , while patients in the Usual Care arm will receive care as usual, and patients in the Neutral Video arm will watch an infant safety video. All measures will be taken in the same way as at the one-month Well Baby visit.

At their four-month Well Baby visit, patients in the TMW-Well Baby arm will watch the Module 3 video intervention , while patients in the Usual Care arm will receive care as usual, and patients in the Neutral Video arm will watch an infant safety video. All measures will be taken in exactly the same way as at the one-month Well Baby visit.

At their six-month Well Baby visit, patients in the TMW-Well Baby arms will watch the Module 4 video intervention, while patients in the Usual Care arm will receive care as usual, and patients in the Neutral Video arm will watch an infant safety video. After the visit, patients in each group will be asked to complete the Post-Visit survey about their appointment. Additional measures will be taken at this visit. The SPEAK will be administered for a second time, the Verbal Comprehension section of the Woodcock-Johnson Test of Cognitive Abilities assessment will be completed, and the participants will be asked to carry out an NCAST PCI teaching task, which is a measure for assessing parent-child interaction via scalable teaching tasks that parents teach their children. Finally, the depression scale results will be shared by the patient's pediatrician, as well as the Ages and Stages Questionnaire (ASQ), if applicable. The Ages and Stages Questionnaire is a screening questionnaire that pinpoints developmental progress in children between the ages of one month to 5 years.

At age seven-months, or about one month after their six-month Well Baby visit, participants will be emailed two follow-up surveys (i.e. the SPEAK and TOPSE surveys). If they complete these surveys within four weeks of receipt, they are eligible for a $10 gift card to be emailed. If the surveys are not completed, participants will not receive the gift-card and will complete these surveys at their next Well-Baby visit.

At their nine-month Well Baby visit, all patients will participate in a second NCAST PCI teaching scale task with their child. At this visit, the MacArthur-Bates Communicative Development Inventories: Words and Gestures Infant form for 8- to 18- month olds (MacArthur-CDI) will be administered. Finally, the depression scale and ASQ results will be shared by the patient's pediatrician, if applicable.

At their twelve-month Well Baby visit, all patients complete the Family Life Events, SPEAK and TOPSE surveys again. Participants will also participate in a third NCAST PCI teaching scale task with their child. The MacArthur-Bates Communicative Development Inventories: Words and Gestures Infant form for 8- to 18- month olds (MacArthur-CDI) will be administered. Finally, any depression scale and ASQ results will be shared by the patient's pediatrician, if applicable.

For participants enrolled on or before 7/31/2016:

At their 18-month Well Baby visit, participants enrolled on or before 7/31/2016 will complete the MacArthur-Bates Communicative Development Inventories Short Form Vocabulary Checklist: Level 1 (MacArthur-CDI) and the SPEAK-R. Finally, any depression scale and ASQ results will be shared by the patient's pediatrician, if applicable.

At their 24-month Well Baby visit, participants enrolled on or before 7/31/2016 will complete the MacArthur-Bates Communicative Development Inventories Short Form Vocabulary Checklist: Level 1 (MacArthur-CDI) and the SPEAK-R. Finally, any depression scale and ASQ results will be shared by the patient's pediatrician, if applicable.

Around age 30-months, participants enrolled on or before 7/31/2016 will be asked to extend their participation in the study to a 30-month home visit and complete the Receptive One-word Picture Vocabulary Test (ROWPVT), Child Behavior Checklist (CBCL), and the Pearlin Mastery Scale.

For participants enrolled between 8/1/2016-1/31/2017:

At their 18-month Well Baby visit, participants enrolled on or before 7/31/2016 will complete the MacArthur-Bates Communicative Development Inventories Short Form Vocabulary Checklist: Level 1 (MacArthur-CDI) and the SPEAK-R. Finally, any depression scale and ASQ results will be shared by the patient's pediatrician, if applicable.

Around age 30-months, participants enrolled between 8/1/2016-1/31/2017, will be asked to extend their participation in the study to a 30-month home visit and participants will complete the Receptive One-word Picture Vocabulary Test (ROWPVT), Child Behavior Checklist (CBCL) , the TOPSE, a survey about seeking advice about child development, and the Pearlin Mastery Scale.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria is as follows: 1) participants (i.e. parents and their children) who live at or below 200% of the federal poverty line, 2) parents at least the age of 18, 3) children younger than 1 month old (at start of study), 4) parents who have legal custody of their child, 5) parents whose child lives with them, 6) parents who are able to commit to the intervention requirements, 7) children who have not experienced any of the following conditions: premature birth (36 weeks or less), cleft lip or cleft palate (and syndromes associated with clefts), Neurocutaneous syndromes (nf1 and 2, tuberous sclerosis, etc), Trisomy, cerebral palsy, history of failing a hearing test, syndromes associated with sensorineural hearing loss (alport, jervell-lange-nielsen, waardenburg, treacher-collins, etc), TORCH infection, Head bleeds or history of intraventricular hemorrhage (IVH), or has had a tracheal intubation, 8) parents who have not earned or are not currently working toward a graduate or professional degree (e.g. M.A., M.S., M.B.A).

Exclusion Criteria:

* 1) participants (i.e. parents and their children) who live over 200% of the federal poverty line, 2) parents under the age of 18, 3) children older than 1 month old (at start of study), 4) parents who do not have legal custody of their child, 5) parents whose child does not live with them, 6) parents who are unable to commit to the intervention requirements, 7) foster parents, 8) children who have experienced any of the following conditions: premature birth (36 weeks or less), cleft lip or cleft palate (and syndromes associated with clefts), Neurocutaneous syndromes (nf1 and 2, tuberous sclerosis, etc), Trisomy, cerebral palsy, history of failing a hearing test, syndromes associated with sensorineural hearing loss (alport, jervell-lange-nielsen, waardenburg, treacher-collins, etc), TORCH infection, Head bleeds or history of intraventricular hemorrhage (IVH), or has had a tracheal intubation, 9) parents who have earned or are currently working toward a graduate or professional degree (e.g. M.A., M.S., M.B.A).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 952 (Actual)
Dates: Start 2016-06; Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
SPEAK | 24 months
  The Survey of Parental Expectations And Knowledge About Language Learning (SPEAK) measures parental knowledge and expectations of how their children learn language at different ages. Some items about beliefs of appropriate age of exposure are rated on a 6-point scale ranging from: 1 "As an infant (0 to 6 moths)" to 6 "In elementary school (6 years and up)" Other items are rated on a 4-point Likert scale ranging from 1 (definitely true), 2 (probably true), 3 (probably not true) to 4 (definitely not true). Scores range from 0 to 71, and scoring of each item is based a criterion scale, with 0 points given to the most incorrect response and 1 additional point given to each progressively more correct response. A higher score correlates to a better outcome and indicates a higher parental knowledge.
Receptive vocabulary score | 30 months
  score of Receptive vocabulary
NCSAT Teaching Scale | 24 months
  Observational data on parent-child interaction. The NCAST Teaching Scale is an assessment for measuring parent-child interaction, and it has 73 variables, which are used to rate caregiver and infant behavior from birth to 36 months. The teaching scale is constructed of 73 item subskills for interaction and marked either yes (1) or no (0) as observed by the clinician during the interaction. The subskills are divided into four subscales for the parent- Sensitivity to Cues, Response to Distress, Social Emotional Growth Fostering, and Cognitive Growth Fostering, and two subscales for the infant-Clarity of Cues and Responsiveness to Caregiver. Summary scores include the total scores for each subscale, the Parent Total Score, Child Total Score, and Parent/Child Total Teaching Score.
Patient report | 24 months
  consistent anticipatory guidance
Stakeholder report | 24 months
  daily anticipatory guidance
TOPSE | 24 months
  Parental self-efficacy measure. The Tool to measure Parenting Self-Efficacy (0-6 months) and can be used to evaluate the effectiveness of parenting programs and identify areas that individual parents may be struggling with. Each statement is scored from 0-10, where 0 equates with "completely disagree," 5 equates with "moderately agree," and 10 equates with "completely agree." Each statement is scored from 0-10 and the total score for each section is a sum of scores. There are 6 sections with 6 questions, including emotion and affection, play and enjoyment, empathy and understanding, pressures, self-acceptance, and learning and knowledge. The booklet comprises of 36 statements in total. The maximum score for each area is 60 and the maximum total score is 360. Higher scores represent a better score.
MacArthur-Bates Communicative Development Inventory (CDI) Vocabulary Checklist: Level 1 | 24 months
  parent report of child's developing abilities in early language
StimQ Cognitive Home Environment | 24 months
  A standardized, interview-based instrument to measure a family's cognitive home environment.
TOI: Survey of Theories of Intelligence | 18 months
  Theories of Intelligence (TOI), which assesses parents' theories about children's intelligence. This 8-item questionnaire measures parents beliefs about the malleability of their child's intelligence. Each question is scored on a likert scale of Strongly Disagree (5) to Strongly Agree (0), with a maximum score of 40. A higher score indicates a better outcome, as it indicates that parents believe that their child's intelligence is malleable.
WJ-IV: Woodcock-Johnson IV Test of Cognitive Abilities: Verbal Reasoning Assessment | 6 months
  The Woodcock Johnson (WJ) assesses a child's school readiness. It measures cognitive abilities, scholastic aptitude, and performance in the areas of reading, mathematics, and written language
CBCL: Child Behavior Checklist | 30 months
  A parent-report questionnaire on which the child was rated on various behavioral and emotional problems. The Child Behavioral Checklist is a checklist assessing concerning and/or troublesome behaviors of children. The CBCL contains 100 items and 3 additional lines of optional items scored from 0-2, with 0 meaning "Not True," 1 meaning "Somewhat or Sometimes True," and 2 meaning "Very true or Often True." The maximum score is 306 (range from 0-306), and higher scores correspond to worse behavior or worse outcomes.

SECONDARY OUTCOMES:
FLE: Family Life Events Survey of family structure, the household, and the child's caretaker(s) | 18 months
  Questionnaire detailing the family structure of the household and the child's caregivers. The Family Life Events Survey (FLE) is a 22-item questionnaire asking about time intensive/potentially stressful family related events in a participants life. Each questions is followed by the answer choices yes (1) or no (0). The maximum score on the survey is 22, and higher scores correspond with more stressful, worse outcomes in terms of stress and family life events.
SDoH: Social Determinants of Health survey | 24 months
  A survey about social determinants of health. The Social Determinants of Health Survey (SDoH) asks questions to help assessor better understand social circumstances that may cause hardship and impact health. There are a total of 14 questions answered with a yes (1) or no (0) in 2 parts. Part 1 contains questions 1-8 and has a maximum score of 8 while Part 2 contains questions 9-14 and has a maximum score of 6. The sum, or total score of the two sections has a maximum score of 14, and higher scores compare to worse outcomes.
ACE: Adverse Childhood Experiences survey | 24 months
  A survey about Adverse Childhood Experiences (ACEs), The Adverse Childhood Experiences (ACE) Survey asks about events occurring during a participant's childhood and tests for the degree of adversity during childhood. There are 17 questions, each with answer choices yes (1) or no (0). There are 2 larger subsections, including household dysfunction and abuse. There are 9 questions involving household dysfunction and 8 involving abuse, and the maximum score is 17. A higher score indicates worse outcome.
EPDS: Edinburgh Postnatal Depression Scale (or other standardized depression scale) | 1 month
  standardized depression scale. The Edinburgh Postnatal Depression Scale measures signs and degree of postnatal depression in mothers. There are a total of 10 questions, scored with varying answers from 0-3. There is a maximum score of 30, which corresponds to higher levels of postnatal depressions and worse outcomes.
ASQ: Ages and Stages Questionnaire | 24 months
  The Ages & Stages Questionnaire: Social-Emotional is a series of questions that aims to identify any social or emotional problems in a developing child.
Pearlin Mastery Scale | 30 months
  The Pearlin Mastery (PM) scale measures the extent to which an individual regards their life chances as being under their personal control rather than fatalistically ruled. The Pearlin Mastery Scale gages how strongly a participant feels that they are able to master and control their lives. There are a total of 7 statements that participants can rate from 1-4 in terms of agreement, where 1 is "Strongly Disagree," 2 is "Disagree," 3 is "Agree," and 4 is "Strongly Agree." The maximum score is 28, and the minimum is 7. A higher score corresponds to higher levels of mastery, or better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Dana Suskind, MD, Principal Investigator — University of Chicago; Kristin Leffel, AB, Study Chair — University of Chicago
Locations (8):
- United States (8):
  - PCC South Family Health Center, Berwyn, Illinois
  - Advocate Medical Group, Chicago, Illinois
  - Lawndale Christian Health Center, Chicago, Illinois
  - University of Chicago Medical Center - Friend Family Health Center, Chicago, Illinois
  - Lawndale Christian Health Center - Archer Avenue, Chicago, Illinois
  - PCC Salud Family Health Center, Chicago, Illinois
  - PCC Austin Family Health Center, Chicago, Illinois
  - PCC Lake Street Family Health Center, Oak Park, Illinois

REFERENCES:
- [Derived] Leung CYY, Trinidad JE, Suskind DL. Video-Based Anticipatory Guidance on Early Cognitive and Language Development in the First 6 Months: A Randomized Controlled Trial. J Pediatr. 2022 Jun;245:227-229.e1. doi: 10.1016/j.jpeds.2022.03.008. Epub 2022 Mar 14. PMID 35301018
- [Derived] List JA, Pernaudet J, Suskind DL. Shifting parental beliefs about child development to foster parental investments and improve school readiness outcomes. Nat Commun. 2021 Oct 1;12(1):5765. doi: 10.1038/s41467-021-25964-y. PMID 34599167
- See also: Click here for more information about the Thirty Million Words — https://tmwcenter.uchicago.edu/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-01): https://cdn.clinicaltrials.gov/large-docs/17/NCT02812017/Prot_SAP_001.pdf